CLINICAL TRIAL: NCT00840008
Title: The Dissemination of Consensus Recommendations on the Management of Canadian Patients With Non Variceal Upper Gastrointestinal Bleeding: A National Cluster Randomized Trial of a Multifaceted Tailored Implementation Strategy
Brief Title: The Dissemination of Consensus Recommendations on Upper Gastrointestinal Bleeding
Acronym: REASON-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Horizon Health Network (Other); Queen Elizabeth II Health Sciences Centre (Other); St-Johns Health Sciences Centre (Unknown); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Jewish General Hospital (Other); Montreal General Hospital (Other); Royal Victoria Hospital, Canada (Other); Maisonneuve-Rosemont Hospital (Other); St Mary's Hospital, London (Other); Centre Hospitalier Pierre Boucher (Unknown); Cité de la Santé Hospital (Unknown); Centre Hospitalier Anna Laberge (Unknown); Hotel Dieu Hospital (Other); CHAUQ - Hopital Saint Sacrement and Hopital Enfant Jesus (Unknown); CISSS de Chaudière-Appalaches (Other Government); Hamilton Health Sciences Corporation (Other); Unity Health Toronto (Other); Sunnybrook Health Sciences Centre (Other); Toronto General Hospital (Other); York Central Hospital, Ontario (Other); Lakeridge Health Corporation (Other); Guelph General Hospital (Unknown); London Health Sciences Centre (Other); The Ottawa Hospital (Other); Kingston Health Sciences Centre (Other); Scarborough General Hospital (Other); Matsqui-Sumas-Abbotsford General Hospital and Mission Memorial Hospital (Unknown); Vancouver General Hospital (Other); Peter Lougheed Centre (Other); Foothills Medical Centre (Other); Alberta Health services (Other); Grey Nuns Hospital (Unknown); University of Alberta (Other); Royal Alexandra Hospital (Other); Misericordia (Unknown); Royal University Hospital Foundation (Other); Regina General Hospital (Other); University of Manitoba (Other)
Responsible Party: Principal Investigator, Alan Barkun, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MCT-88113
Record Dates: First submitted 2009-02-04; First posted 2009-02-10 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: peptic ulcer bleeding; upper GI hemorrhage; adherence to guidelines; knowledge transfer
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Gastrointestinal Hemorrhage | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational intervention (Experimental): see protocol
  Interventions: Other: Educational intervention
- Standard care (No Intervention): distribution of guidelines and a published algorithm

INTERVENTIONS:
Other: Educational intervention — As per detailed protocol.
  Other Names: Multifacetted tailored educational intervention
  Arms: Educational intervention

SUMMARY:
The purpose of this study is to assess whether adherence to NVUGIB guidelines is improved with implementation of a national, tailored multifaceted intervention. Outcomes include adherence rates to two key endoscopic and pharmacological therapy guidelines together (primary), or adherence to these individually as well as to other recommendations (secondary). Patient outcomes and economic data are also assessed (tertiary).

DETAILED DESCRIPTION:
Clusters are randomized to receive a published algorithm and guidelines (control group), or a multifaceted, tailored educational intervention (see details in protocol - intervention group). The charts of treated patients with non variceal upper GI bleeding are reviewed and adherence to selected guidelines recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over.
* Treated during the study duration
* Primary or secondary discharge diagnoses of NVUGIB (per charted ICD-10 code). Additional confirmation of NVUGIB using endoscopic findings or patient symptoms done as previous.

Exclusion Criteria:

* Patients initially assessed at another institution for the present episode of NVUGIB and subsequently transferred to the participating site with unavailable initial data.
* Endoscopy noted no gastro-duodenal ulcer bleeding, to ensure patient homogeneity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3157 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adherence to guidelines G10 and G17 of the 2003 International Consensus Guidelines on nonvariceal upper GI bleeding. | 1 year

SECONDARY OUTCOMES:
Adherence to guidelines G10 or G17 alone, G5b, G6, G7a, G7b , G7c, G18 of the 2003 International Consensus Conference on nonvariceal upper GI bleeding. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alan Barkun, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre

REFERENCES:
- [Derived] Barkun AN, Bhat M, Armstrong D, Dawes M, Donner A, Enns R, Martin J, Moayyedi P, Romagnuolo J, Stitt L. Effectiveness of disseminating consensus management recommendations for ulcer bleeding: a cluster randomized trial. CMAJ. 2013 Feb 19;185(3):E156-66. doi: 10.1503/cmaj.120095. Epub 2013 Jan 14. PMID 23318399